CLINICAL TRIAL: NCT04572906
Title: Phase 2a, Multicenter, Randomized, Patient and Evaluator Blinded, Controlled Study Evaluating the Safety and Efficacy of NTX-001 Compared to SOC in the Treatment of Acute Single Transected Peripheral Nerve Injury Occurring Below the Distal Border of the Brachial Plexus Requiring Surgical Repair.
Brief Title: Safety and Efficacy of NTX-001 Compared to SOC in Acute Single Peripheral Nerve Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuraptive Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTx20201
Record Dates: First submitted 2020-09-10; First posted 2020-10-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Treatment vs. Standard of Care
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All study personnel involved in the surgical procedure will be unblinded. Patient and outcomes evaluators will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NTX-001 (Experimental): NTX-001 used during surgical repair of an upper extremity peripheral nerve injury in conjuction with standard suture neurorrhaphy.
  Interventions: Combination Product: NTX-001
- Standard of Care (No Intervention): standard suture neurorrhaphy

INTERVENTIONS:
Combination Product: NTX-001 — One time use surgical product, 3 solutions applied topically, in sequence, to the peripheral nerve repair site, in conjunction with standard suture neurorrhaphy. An isolation chamber medical device (device) is utilized to focus the application of PEG (Solution #2) on the coapted nerve for the required amount of exposure time.
  Other Names: PEG-fusion
  Arms: NTX-001

SUMMARY:
NTX-001 is a single use surgical product intended for use in conjunction with standard suture neurorrhaphy of severed nerves in patients between 16 and 80 years of age.

DETAILED DESCRIPTION:
NTX-001 (Product) is a surgical product that consists of an active solution (drug), an isolation chamber medical device (chamber or device) and two (2) other sterile solutions.

NTX-001 has been developed as a surgical product to be used in conjunction with standard suture neurorrhaphy of a severed nerve. Use of NTX-001 is intended to safely accelerate the often slow and diminished return of function in repaired nerves. It often takes months and/or years to determine if function will be restored. By that point, restoration is often incomplete and can result in lifelong motor and/or sensory deficits. By reconnecting (PEG-fusion) a substantial number of axons within a severed nerve, the degeneration-regeneration cycle and subsequent atrophy may be reduced or even prevented for those axons and their targets, respectively. NTX-001 (PEG-fusion) has the potential to avoid the consequences of protracted denervation of distal target tissues by eliminating the period of total denervation thus reducing the time to stable recovery and providing greater innervation to affected tissues.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 12 years of age and not older than 80.
* The subject has sustained a confirmed (intra-op assessment) single transected peripheral nerve injury.
* The subject's nerve injury is classified as Sunderland's Fourth and Fifth Degree (Class III)
* The subject's nerve injury is amenable to minimal or acceptable tension, in direct, end-to-end repair.
* The surgical repair will occur within 48 hours of injury.

Exclusion Criteria:

* The subject has a PNI with a segmental loss (gap) that cannot be repaired with minimal or acceptable tension.
* Other treatments known to affect the growth and/or physiology of the neural and vascular system.
* The nerve injury has vascular damage that cannot be repaired to provide adequate perfusion of the injured site.
* The subject is pregnant and/or is breastfeeding.
* The subject has a significant medical comorbidity precluding immediate repair.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events | Up to 48 Weeks
  An adverse event is any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given a study product or in a clinical study. A treatment-emergent adverse event was defined as any adverse event that newly appeared, increased in frequency, or worsened in severity on or after the exposure to the study product.
Michigan Hand Questionnaire Total Score (MHQ) | Week 12
  The MHQ measures hand function and is scored from 0-100; with 100 being the "best" score.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Weeks 4, 8, 12, 24, 36 and 48
  The NPRS measures pain intensity on a scale from 0 representing no pain and 10 to the worst pain as bad as you can imagine.
Modified British Medical Research Council (MMRC) sensory grading (S0-S4) | Weeks 4, 8, 12, 24, 36 and 48
  The SWMT measures sensation as using a score from S0 to S4; higher score indicates better sensation.
Modified British Medical Research Council (MMRC) motor grading (M0-M5) | Weeks 4, 8, 12, 24, 36 and 48
  The MRCC motor measures the function of the muscles; on a scale from M0 to M5; the higher score indicates better strength.
Semmes-Weinstein Monofilament Test (SWMT) | Weeks 4, 8, 12, 24, 36 and 48
  The SWMT assesses sensation using using equipment that measures force felt in grams.
Pinch Strength | Weeks 4, 8, 12, 24, 36 and 48
  The Pinch test assesses strength using using equipment that measures strength in pounds.
Grip Strength | Weeks 4, 8, 12, 24, 36 and 48
  The Grip test assesses strength using using equipment that measures strength in pounds.
Cold Intolerance Symptom Severity (CISS) | Weeks 4, 8, 12, 24 and 48
  The CISS focuses on the impact of cold intolerance on activities of daily life; the score ranges a score between 0 and 10, where 0 is no symptoms at all and 100 is the most severe symptoms you can possibly imagine.
Patient Global Impression of Change (PGIC) | Weeks 4, 8, 12, 24 and 48
  The PGIC measures information about the effect of a treatment intervention in an individual subject, scored 0 to 7; with 0 being the worst and 7 being the best.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Schulman, MD, Study Chair — Neuraptive Therapeutics Inc.
Locations (10):
- United States (10):
  - UF Health - University of FL - Gainesville, Gainesville, Florida
  - Orlando Health, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - Curtis National Hand Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - The Ohio State University Wexner Medical Center Hand and Upper Extremity Center, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghergherehchi CL, Mikesh M, Sengelaub DR, Jackson DM, Smith T, Nguyen J, Shores JT, Bittner GD. Polyethylene glycol (PEG) and other bioactive solutions with neurorrhaphy for rapid and dramatic repair of peripheral nerve lesions by PEG-fusion. J Neurosci Methods. 2019 Feb 15;314:1-12. doi: 10.1016/j.jneumeth.2018.12.015. Epub 2018 Dec 23. PMID 30586569
- [Background] Mikesh M, Ghergherehchi CL, Louis Hastings R, Ali A, Rahesh S, Jagannath K, Sengelaub DR, Trevino RC, Jackson DM, Bittner GD. Corrigendum to "Polyethylene glycol solutions rapidly restore and maintain axonal continuity, neuromuscular structures, and behaviors lost after sciatic nerve transections in female rats.". J Neurosci Res. 2018 Sep;96(9):1623. doi: 10.1002/jnr.24277. No abstract available. PMID 30113719
- [Background] Mikesh M, Ghergherehchi CL, Rahesh S, Jagannath K, Ali A, Sengelaub DR, Trevino RC, Jackson DM, Tucker HO, Bittner GD. Corrigendum to "Polyethylene glycol treated allografts not tissue matched nor immunosuppressed rapidly repair sciatic nerve gaps, maintain neuromuscular functions, and restore voluntary behaviors in female rats". J Neurosci Res. 2018 Sep;96(9):1624. doi: 10.1002/jnr.24278. No abstract available. PMID 30113723
- [Background] Bittner GD, Spaeth CS, Poon AD, Burgess ZS, McGill CH. Repair of traumatic plasmalemmal damage to neurons and other eukaryotic cells. Neural Regen Res. 2016 Jul;11(7):1033-42. doi: 10.4103/1673-5374.187019. PMID 27630671
- [Background] Bittner GD, Sengelaub DR, Trevino RC, Peduzzi JD, Mikesh M, Ghergherehchi CL, Schallert T, Thayer WP. The curious ability of polyethylene glycol fusion technologies to restore lost behaviors after nerve severance. J Neurosci Res. 2016 Mar;94(3):207-30. doi: 10.1002/jnr.23685. Epub 2015 Nov 3. PMID 26525605